CLINICAL TRIAL: NCT00308932
Title: Relative Amount of Fluticasone Delivered by HFA-MDI Through Chamber/Mask to Young Children With Asthma
Brief Title: Effect of Age and Device on Delivery of Fluticasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38-2002
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2004-08

CONDITIONS: Asthma
Keywords: fluticasone; asthma therapy; spacer inhaler; HFA-134a
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: HFA FP MDI

SUMMARY:
To determine the effect of age and device on delivery of HFA-Fluticasone Propionate (FP) in children of different ages. Hypothesis -- passive inhalation in younger children through a valved holding chamber/mask (VHC) will reduce the relative amount of FP delivered to airways.

DETAILED DESCRIPTION:
The objective was to determine the effect of age and device on delivery of fluticasone propionate delivered by HFA-pMDI in children of different ages. The one-hour steady-state fluticasone plasma concentration which is an indirect measure of airway delivery and direct measure of systemic exposure, was determined. Sixty children with well-controlled persistent asthma received two actuations of 110 mcg twice daily for at least 3 days. A blood sample was collected one hour after the last dose when 100% adherence was documented by electronic monitor. Five groups of 12 each were studied: 1) 12-18 yr by actuator alone; 2) 5-9 yr by actuator alone; 3) 5-9 yr by antistatic VHC/mouthpiece; 4) 5-9 yr by antistatic VHC/mask and 5) 1-4 yr by antistatic VHC/mask. Fluticasone concentrations were measured by LC-MS/MS assay. Fluticasone plasma concentration between groups was compared using one way ANOVA.

ELIGIBILITY:
Inclusion Criteria:children 1-18 yr, adequately controlled persistent asthma, demonstrate effective administration technique in accordance with the group assigned -

Exclusion Criteria:inadequately controlled asthma: nocturnal awakening >2 nights/month, prn albuterol use >2x/week, more than 2 short courses of oral corticosteroids in previous 3 months, missing a dose on more than one occasion, increase in asthma symptoms during study, inability to discontinue intranasal or dermal fluticasone for 3 days

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2003-02; Study Completion 2004-04

PRIMARY OUTCOMES:
One-hour steady-state plasma concentration of fluticasone

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hendeles, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Asthma Research Lab, Gainesville, Florida, United States